CLINICAL TRIAL: NCT00673335
Title: Prevention of Breast Cancer by Letrozole in Post-menopausal Women Carrying a BRCA1/BRCA2 Mutation
Brief Title: Letrozole in Preventing Breast Cancer in Postmenopausal Women With a BRCA1 or BRCA2 Mutation
Acronym: LIBER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UC-0104/0701 - ONCO03; ONCO-03/0701 (Other: UNICANCER); EU-20806; NOVARTIS-FNCLCC-ONCO 03/0701; 2007-000687-24 (EudraCT Number)
Record Dates: First submitted 2008-05-06; First posted 2008-05-07 (Estimated); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: brca1 Mutation Carrier; brca2 Mutation Carrier; Breast Cancer; Hereditary Breast/Ovarian Cancer (brca1, brca2)
Keywords: breast cancer; hereditary breast/ovarian cancer (BRCA1, BRCA2); BRCA1 mutation carrier; BRCA2 mutation carrier
MeSH Terms: conditions — Breast Neoplasms; Hereditary Breast and Ovarian Cancer Syndrome | interventions — Letrozole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment arm (Experimental): Letrozole, 1 tablet
  Interventions: Drug: letrozole
- Placebo (Placebo Comparator): Comparator, 1 tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: letrozole
  Other Names: Femara
  Arms: Treatment arm
Drug: Placebo
  Arms: Placebo

SUMMARY:
RATIONALE: Letrozole may prevent breast cancer in postmenopausal women with a BRCA1 or BRCA2 mutation.

PURPOSE: This randomized phase III trial is studying letrozole to see how well it works compared with a placebo in preventing breast cancer in postmenopausal women with a BRCA1 or BRCA2 mutation.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the reduction of the incidence of invasive breast cancer in postmenopausal women with the BRCA1/BRCA2 mutation treated with letrozole.

Secondary

* Determine the reduction of the incidence of in situ breast cancer in these women.
* Determine the recurrence rate of local or metastatic disease in women who have had breast cancer.
* Determine the incidence of non-breast cancer, especially ovarian, colon, or endometrial cancer.
* Assess the tolerance of this drug in terms of lipid, cardiovascular, and bone effects.
* Determine the quality of life of women treated with this drug.
* Identify serological markers that allow early diagnosis of hereditary predisposition for breast cancer.
* Conduct pharmacogenetic analysis.
* Identify biomarkers or genes involved in the occurrence of cardiovascular and rheumatologic metabolic aromatase inhibitors.
* Study the phenotypic characteristics of cancers that occur during treatment with letrozole, in particular hormonal markers (estrogen and progesterone receptor) and expression profiles of resistance to therapy.

OUTLINE: This is a multicenter study. Patients are stratified according to nature of mutation (BRCA1 vs BRCA2), oophorectomy in premenopausal state (yes vs no), and prior breast cancer (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral letrozole once daily.
* Arm II: Patients receive oral placebo once daily. Treatment in both arms continues for 5 years in the absence of unacceptable toxicity or development of cancer or recurrent disease.

Blood samples are collected periodically for pharmacogenetic studies and analysis of biomarkers or genes associated with hereditary predisposition for breast cancer, toxicities, and resistance to therapy.

After completion of study treatment, patients are followed for 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Must meet the following criteria:

  * With or without invasive unilateral breast cancer more than 5 years ago, with no recurrence

    * No evidence of breast cancer by mammography or MRI within the past year
  * Carrier of the BRCA1/BRCA2 deleterious mutation (nonsense mutation or stop)
  * Refused preventive mastectomy
* No prior bilateral breast cancer
* No prior bilateral mastectomy
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

Inclusion criteria:

* Menopausal status as indicated by 1 of the following criteria:

  * Age > 60 years
  * Bilateral oophorectomy
  * Age ≤ 60 years with no hysterectomy or amenorrhea within the past 12 months
  * Age ≤ 60 years with prior hysterectomy or FSH > 20 IU/L
* Eastern Cooperative Oncology Group (ECOG) or WHO performance status 0-1
* absolute neutrophil count (ANC) > 2,000/mm^3
* Platelet count > 100,000/mm^3
* Hemoglobin > 10 g/dL
* Bilirubin normal
* ALT and AST < 2.5 times upper limit of normal
* Creatinine clearance ≥ 60 mL/min
* Adequate cardiovascular function (e.g., no history of myocardial infarction, angina pectoris, or heart failure)
* No osteoporosis by bone density scan (DEXA) within the past 2 years or prior osteoporotic fracture (femur, lumbar spine T score > -2 DS)

Exclusion criteria:

* Invasive cancer diagnosed in the past 5 years, except for basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* Prior cerebrovascular accident
* Prior cardiac ischemia
* Hypersensitivity to letrozole or its excipients, especially titanium oxide
* Renal or hepatocellular insufficiency, cholestasis, or cytolysis
* Geographical, social, or psychological reasons that preclude medical monitoring in this study
* Deprived of liberty or guardianship

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 3 months since prior and no concurrent hormone replacement therapy (e.g., thyroid-stimulating hormone)
* No prior hormonal therapy in the past year
* No concurrent participation in another therapeutic study with an experimental drug

Ages: 40 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2008-05 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2023-12 (Actual)

PRIMARY OUTCOMES:
Survival without contralateral or unilateral invasive breast cancer at 5 years (prior breast cancer) | 2017
Survival without invasive breast cancer at 5 years | 2017

SECONDARY OUTCOMES:
Invasive cancer-free survival at 10 years | 2022
Breast cancer in situ-free survival at 5 and 10 years | 2022
Relapse-free (local or metastatic disease) survival in patients with history of breast cancer at 5 and 10 years | 2017 and 2022
Second cancer-free survival at 5 and 10 years | 2017 and 2022
Event- free (local relapse or metastatic, contralateral, or second cancer) survival at 5 and 10 years | 2017 and 2022
Overall survival at 5 and 10 years | 2017 and 2022
Toxicity according to CTCAE version 3.0 | 2017 and 2022
Lipid tolerance or cardiovascular or bone event | 2017 and 2022
Quality of life according to MRS and SF36 questionnaires | 2017 and 2022

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Pujol, MD, Study Chair — Hopital Arnaud de Villeneuve
Locations (23):
- France (23):
  - Institut Sainte Catherine, Avignon
  - Centre Regional Francois Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Marseille Institute of Cancer - Institut J. Paoli and I. Calmettes, Marseille
  - Hopital Arnaud de Villeneuve, Montpellier
  - Centre Catherine de Sienne, Nantes
  - Centre Antoine Lacassagne, Nice
  - Centre Hospitalier General de Niort, Niort
  - Hopital Saint Michel, Paris
  - Hotel Dieu de Paris, Paris
  - Institut Curie Hopital, Paris
  - CHU Poitiers, Poitiers
  - Polyclinique De Courlancy, Reims
  - Centre Eugene Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - Centre Rene Huguenin, Saint-Cloud
  - CHU Sainte-Etienne - Hopital Nord, Saint-Etienne
  - Centre Paul Strauss, Strasbourg
  - Institut Claudius Regaud, Toulouse
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Yes
Unicancer will share de-identified individual data that underlie the results reported. A decision concerning the sharing of other study documents, including protocol and statistical analysis plan will be examined upon request.
Supporting Information: Study Protocol, SAP
Time Frame: Unicancer will consider access to study data upon written detailed request sent to Unicancer, from 6 months until 5 years after publication of summary data.
Access Criteria: The data shared will be limit to that required for independent mandated verification of the published results, the applicant will need authorization from Unicancer for personal access, and data will only be transferred after signing of a data access agreement.

REFERENCES:
- [Background] Pujol P, Lasset C, Berthet P, Dugast C, Delaloge S, Fricker JP, Tennevet I, Chabbert-Buffet N, This P, Baudry K, Lemonnier J, Roca L, Mijonnet S, Gesta P, Chiesa J, Dreyfus H, Vennin P, Delnatte C, Bignon YJ, Lortholary A, Prieur F, Gladieff L, Lesur A, Clough KB, Nogues C, Martin AL; French Federation of Cancer Centres (FNCLCC). Uptake of a randomized breast cancer prevention trial comparing letrozole to placebo in BRCA1/2 mutations carriers: the LIBER trial. Fam Cancer. 2012 Mar;11(1):77-84. doi: 10.1007/s10689-011-9484-4. PMID 22076253
- [Result] Pujol P, Mijonnet S, Karen S, et al.: Breast cancer prevention by letrozole in post menopausal BRCA1/2 mutations carriers: The Onco-03/LIBER trial. [Abstract] 32nd Annual San Antonio Breast Cancer Symposium, December 9-13, 2009, San Antonio, Texas. A-1048, 2009.